CLINICAL TRIAL: NCT03892746
Title: Improving SCI Rehabilitation Interventions by Retraining the Brain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ela B. Plow, Principal Investigator, Staff, Neural Control Lab, Dept. of Biomedical Engineering, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-972; CDMRP-SC170311 (Other Grant/Funding Number: Congressionally Directed Medical Research Program Program (CDMRP), DoD)
Record Dates: First submitted 2019-01-17; First posted 2019-03-27 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Cervical Spinal Cord Injruy
Keywords: Cervical Spinal Cord Injury; tDCS; Transcranial Direct Current Stimulation; Upper limb; Rehabilitation; Brain Stimulation

STUDY DESIGN:
Intervention Model Description: In this phase I/II clinical trial, an anticipated 49(up to 54) subjects will receive 15 sessions of upper limb training while receiving either active tDCS or sham tDCS to the target in the brain devoted to the weaker triceps of the weaker upper limb.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomly assigned by the Cleveland Clinic biostatistician to receive either active or sham tDCS. The tDCS will be pre-programmed with codes for active and sham stimulation. The code will be given to the intervention team by the biostatistician. Investigators analyzing functional outcome data and neurophysiology data will receive coded data that conceals the identity of the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active tDCS + task oriented practice (Active Comparator)
  Interventions: Device: Active tDCS + task oriented practice
- Sham tDCS + task oriented practice (Sham Comparator)
  Interventions: Device: Sham tDCS + task oriented practice

INTERVENTIONS:
Device: Active tDCS + task oriented practice — Participants in this arm will receive active tDCS (2mA) to the motor cortex (targeting the triceps) of the weaker upper limb for 2, 30-minute cycles during each 2-hour upper limb training session. While receiving tDCS, the participant will be performing task-oriented practice for the weaker upper limb. Participants will receive these interventions for 15 sessions over several weeks up to 8 weeks.
  Arms: Active tDCS + task oriented practice
Device: Sham tDCS + task oriented practice — Participants in this arm will receive sham tDCS (0mA) to the motor cortex (targeting the triceps) of the weaker upper limb for 2, 30-minute cycles during each 2-hour upper limb training session. While receiving tDCS, the participant will be performing task-oriented practice for the weaker upper limb. Participants will receive these interventions for 15 sessions over several weeks up to 8 weeks.
  Arms: Sham tDCS + task oriented practice

SUMMARY:
The Long-term goal of this project is to develop upper limb rehabilitation interventions that can be utilized for cervical Spinal Cord Injury survivors.

This Study will utilize a novel method of non-invasive brain stimulation in conjunction with upper limb training given for 15 sessions over several weeks up to 8 weeks.

The Study will include the following site visits:

* Eligibility Screening and Informed Consent Visit.
* Four testing visit in which motor function of the upper limb and neurophysiology will be measured
* Fifteen intervention visits during which patients will receive upper limb training in conjunction with non-invasive brain stimulation
* Repeat testing of motor function and neurophysiology of the upper limb following completion of intervention visits
* a Follow-up visit completed 3 months after the completion of interventions

DETAILED DESCRIPTION:
This is a phase I/II Multi-site Clinical Trial. In this phase I/II randomized controlled study, 49(up to 54) cervical spinal patients with upper limb impairments will receive non-invasive brain stimulation tDCS (Transcranial Direct Current Stimulation) to the area in the brain controlling the weaker muscle of the weakest upper limb while receiving training for 15 sessions over several weeks up to 8 weeks. The primary outcome will be motor limb impairment, and secondary outcomes will be tests of functional ability, spinal excitability, and strength and dexterity. Safety and feasibility of pairing tDCS with rehabilitation will also be explored and include adverse effects, subject/investigator blinding, and attrition to 3 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with incomplete (having sparing to muscles in the upper extremities below the level of injury) C1-C8 SCI
* at least 1 year post injury
* weakness of the triceps or biceps muscle in the weaker upper limb, defined as a clinically detectable difference in power compared to the power of the spared antagonist(biceps and triceps respectively) muscle, i.e., at least one muscle grade lower on the MRC scale.

Exclusion Criteria:

* contraindications to tDCS and TMS including: pacemaker, metal in the skull, seizure history, pregnancy.
* pressure ulcers
* traumatic brain injury (TBI), diagnosed based upon acute injury Rancho scale <5 or positive MRI/CT findings at the time of injury will also be excluded to prevent confounding of TMS metrics.
* excessive tone/spasticity and severe contractures or soft tissue shortening at the elbow/wrist
* participating in ongoing upper-limb therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ela Plow, PhD, Principal Investigator — The Cleveland Clinic
Locations (4):
- United States (4):
  - Kessler Foundation, West Orange, New Jersey
  - Louis B. Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - Lerner Research Institute; Cleveland Clinid Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arora T, O'Laughlin K, Potter-Baker K, Kirshblum S, Kilgore K, Forrest GF, Bryden AM, Wang X, Henzel MK, Li M, Perlic K, Richmond MA, Pundik S, Bethoux F, Frost F, Plow EB. Safety and efficacy of transcranial direct current stimulation in upper extremity rehabilitation after tetraplegia: protocol of a multicenter randomized, clinical trial. Spinal Cord. 2022 Sep;60(9):774-778. doi: 10.1038/s41393-022-00768-z. Epub 2022 Mar 5. PMID 35246620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All spinal cord injury (SCI) participants were enrolled in the study between July 2019 and August 2024. Enrollment sites included the Cleveland Clinic, Louis Stokes Cleveland VA Medical Center, Kessler Institute for Rehabilitation, and MetroHealth Hospital. Following the provision of informed consent, participants underwent an eligibility assessment to confirm study qualifications were met.
Pre-assignment Details: Of the 47 enrolled SCI participants, six were excluded prior to group assignment. Reasons for exclusion include voluntarily withdrawal (5) and unable to proceed due to clinical care requirements (1). The remaining 41 participants were randomized and competed study procedures.
Period: Overall Study
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
Started | 20 | 21
Completed | 16 | 20
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active tDCS + Task Oriented Practice: Active tDCS + task oriented practice: Participants in this arm will receive active tDCS(2mA) to the motor cortex(targeting the triceps) of the weaker upper limb for 2 30 minute cycles during each 2 hour upper limb training session. While receiving tDCS the participant will be performing task oriented practice for the weaker upper limb. Participants will receive these interventions for 15 sessions over several weeks up to 8 weeks.
- Sham tDCS + Task Oriented Practice: Sham tDCS + task oriented practice: Participants in this arm will receive sham tDCS(0mA) to the motor cortex(targeting the triceps) of the weaker upper limb for 2 30 minute cycles during each 2 hour upper limb training session. While receiving tDCS the participant will be performing task oriented practice for the weaker upper limb. Participants will receive these interventions for 15 sessions over several weeks up to 8 weeks
- Total: Total of all reporting groups
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (16) | 48 (17) | 48 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Upper Extremity Motor Score (UEMS) With Manual Muscle Testing
Description: UEMS is used in Spinal Cord injury to identify strength (muscle power) in patients with spinal cord injury. It involves a manual muscle test of five key muscles in each arm graded from 0 (no contraction) to 5 (normal strength). Each Arm can have a max score of 25 and the total score for the test is 50 points. The higher the value the more muscle strength the participant has and a higher change score means more improvement. The sum of scores for both arms is reported here.
Time Frame: Baseline (0 weeks), after intervention (up to 8 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
Number analyzed (Participants) | 16 | 20
score on a scale | 3.5 (0.67) | 2.55 (.67)

2. Primary Outcome: Change in Graded and Redefined Assessment of Strength, Sensibility and Prehension (GRASSP)
Description: Graded and Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) is a functional measure which identifies the functional ability of the upper limbs and is widely used in studies recruiting Spinal Cord Injury patients. It has subsets including strength (100 points total, 50 per arm), palmar and dorsal sensation (48 points total, 24 per arm), prehension ability (24 points total, 12 per arm), and prehension performance (60 points total, 30 per arm). The higher the score the better the performance. The greater the change in score the more the participant improved. The sum of scores for both arms is reported here.
Time Frame: Baseline (0 weeks), after intervention (up to 8 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
Number analyzed (Participants) | 16 | 20
units on a scale | 9.56 (2.96) | 10.3 (1.74)

3. Primary Outcome: Change in Canadian Occupational Performance Measure (COPM) Performance
Description: The Canadian Occupational Performance Measure (COPM) is an evidence-based outcome measure designed to capture the participants self-perception of everyday issues that restrict their participation in everyday living, measuring both their performance in completing the identified task and their satisfaction in their performance of the task. Here we report the performance scale of the assessment. The score range is from minimum 1 (not able to do it at all) and maximum 10 (able to do it extremely well). A larger change score indicates more subjective improvement in performance of activies of daily living.
Time Frame: Baseline (0 weeks), after intervention (up to 8 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
Number analyzed (Participants) | 16 | 20
score on a scale | 0.89 (0.22) | 0.77 (0.33)

4. Primary Outcome: Change in Canadian Occupational Performance Measure (COPM) Satisfaction
Description: The Canadian Occupational Performance Measure (COPM) is an evidence-based outcome measure designed to capture the participants self-perception of everyday issues that restrict their participation in everyday living, measuring both their performance in completing the identified task and their satisfaction in their performance of the task. Here we report the satisfaction scale of the assessment. The score range is from minimum 1 (not satisfied at all) and maximum 10 (extremely satisfied). A larger change score indicates more subjective improvement in satisfaction of completing activies of daily living.
Time Frame: Baseline (0 weeks), after intervention (up to 8 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
Number analyzed (Participants) | 16 | 20
score on a scale | 0.92 (0.25) | 1.36 (0.37)

5. Primary Outcome: Change in Spinal Cord Independence Measure (SCIM), Self-care Subscore
Description: The Spinal Cord Indepence Measure (SCIM) is a participant subjective spinal cord injury measure that identifies daily acitivity indepence. The Self-care subscore of the SCIM looks at independence in performing daily activies and ranges from minimum 0 (total dependence in self-care) to maximum 20 (complete independence in self-care). A higher change score indicates improved levels of independece for the participant.
Time Frame: Baseline (0 weeks), after intervention (up to 8 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
Number analyzed (Participants) | 16 | 20
score on a scale | 0.62 (0.38) | 0.3 (0.44)

6. Primary Outcome: Change in Capabilities of Upper Extremity Test (CUE-T)
Description: The Capabilities of Upper Extremity Test (CUE-T) is a performance based functional measure that evaluates upper extremity function in poeple with cervical spinal cord injury. It consists of 32 items, each item is scored from 0 (unable to complete task) to 4 (no difficulty to complete task). The minimum score of the scale is 0 (unable to performe any of the tasks) to maximum 128 (able to complete every task with no difficulty). A higher change score indicates and improvement in ability to complete upper limb functional tasks.
Time Frame: Baseline (0 weeks), after intervention (up to 8 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
Number analyzed (Participants) | 16 | 20
score on a scale | 3.44 (1.26) | 3.75 (0.93)

7. Primary Outcome: Change in Excitability (Active Motor Threshold) of Cortical and Corticospinal Physiology (TMS), Weaker Arm-Biceps
Description: Transcranial magnetic stimulation was used to test cortical and corticospinal physiology. The active motor threshold (AMT) is the lowest intensity of stimulation needed to produce a motor evoked potential during a voluntary contraction in the biceps muscle. The criteria for defining a motor evoked potential is 6 out of 10 trials in which the response signal is larger peak-to-peak than the background muscle activity by 100µV. The AMT can have a value ranging from 0-100, an indicator of the percentage of the maximum stimulator output (MSO). The higher the value the more stimulation intensity needed to get a criterion motor evoked potential in the target muscle; lower AMT values indicate higher excitability in the muscle. A change score that is negative indicates increased excitability in the biceps muscle.
Time Frame: Baseline (0 weeks) and after intervention (up to 8 weeks)
Population: Three participants (2 active, 1 sham) were excluded from the analysis as they did not complete both pre and post testing due to voluntarily opting out of undergoing the neurophysiology testing session.
Measure: Mean (Standard Error); unit: Percentage of MSO
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
Number analyzed (Participants) | 14 | 19
Percentage of MSO | 1.1 (3.4) | -0.9 (1.1)

8. Primary Outcome: Change in Excitability (Active Motor Threshold) of Cortical and Corticospinal Physiology (TMS), Weaker Arm Triceps
Description: Transcranial magnetic stimulation was used to test cortical and corticospinal physiology. The active motor threshold (AMT) is the lowest intensity of stimulation needed to produce a motor evoked potential during a voluntary contraction in the triceps muscle. The criteria for defining a motor evoked potential is 6 out of 10 trials in which the response signal is larger peak-to-peak than the background muscle activity by 100µV. The AMT can have a value ranging from 0-100, an indicator of the percentage of the maximum stimulator output (MSO). The higher the value, the more stimulation intensity needed to get a criterion motor evoked potential in the target muscle; lower AMT values indicate higher excitability in the muscle. A change score that is negative indicates increased excitability in the triceps muscle.
Time Frame: Baseline (0 weeks) and after intervention (up to 8 weeks)
Population: One participant (1 active) was excluded from the analysis as they did not complete both pre and post testing due to voluntarily opting out of undergoing the neurophysiology testing session.
Measure: Mean (Standard Error); unit: Percentage of MSO
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
Number analyzed (Participants) | 15 | 20
Percentage of MSO | 0.1 (1.1) | -2.2 (2.9)

9. Primary Outcome: Change in Excitability of Spinal Physiology of the Flexor Carpi Radialis Muslce in the Weaker Arm.
Description: Spinal pathways were tested using peripheral nerve stimulation to median nerve to collect responses in the Flexor Carpi Radialis muscle of the weaker arm. This stimulation stimulates both the sensory and motor nerves to produce a evoked potential for each pathway. The evoked potential produced for the sensory pathway is considered the Hoffman reflex (H-reflex) and the evoked potential produced for the motor pathway is considered the muscle compund action potential (M-wave). To get an understanding of the motor neuron pool of exitability we use the H/M ratio which compares the peak amplitude of the maximum H-reflex to the maximum M-wave (H-reflex/M-wave). This ratio reflects the proportion of the motor neruon pool activated by the reflex or motor neuron excitability. A lower H/M ratio generally indicates lower excitability while a higher ratio indicates higher excitability.
Time Frame: Baseline (0 weeks) and after intervention (up to 8 weeks)
Population: Peripheral nerve stimulation in SCI participants can be painful due to heightened sensitivity. Also due to limitations of stimulator output we may not have seen a signal to analyze. Therefore only 6 participants in the active group and 10 participants in the sham group had eligible data to analyze from baseline to post test
Measure: Mean (Standard Error); unit: change in H/M ratio
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
Number analyzed (Participants) | 6 | 10
change in H/M ratio | -5.1 (4.7) | -0.7 (4.5)

10. Other Pre Specified Outcome: Safety and Feasibility
Description: In line with this phase I/II clinical trial, safety and feasibility will be tested throughout this study. Vital signs (blood pressure, heart rate, respirations, blood oxygen saturation) will be recorded for each study session. During Intervention sessions we will ask a tDCS adverse effects questionnaire at the end of each session.
Time Frame: Through study completion, an average of 7 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: TMS Safety Questionnaire
Description: A TMS safety questionnaire will be asked at the end of the preintervention tests and the post intervention testing visit.
Time Frame: Baseline (0 weeks) and after intervention (up to 8 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 7 months
Arm/Group | Active tDCS + Task Oriented Practice | Sham tDCS + Task Oriented Practice
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 16/20 | 15/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active tDCS + Task Oriented Practice (N=20) | Sham tDCS + Task Oriented Practice (N=21)
Redness at Site of Stimulation (Skin and subcutaneous tissue disorders) | 4 | 7
Dizziness (Nervous system disorders) | 0 | 1
Disorientation/Confusion (Nervous system disorders) | 0 | 1
Tingling Sensation (Skin and subcutaneous tissue disorders) | 16 | 15
Itching Sensation (Skin and subcutaneous tissue disorders) | 14 | 10
Burning Sensation (Skin and subcutaneous tissue disorders) | 13 | 14
Pain at the site of stimulation (Skin and subcutaneous tissue disorders) | 3 | 4
Headache (Nervous system disorders) | 6 | 4
Difficulties in concentrating (Nervous system disorders) | 1 | 2
Visual sensations associated with stimulation (Nervous system disorders) | 2 | 0
Nervousness (Social circumstances) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT03892746/Prot_SAP_003.pdf
  • Informed Consent Form (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT03892746/ICF_001.pdf